CLINICAL TRIAL: NCT05072223
Title: Efficacy and Safety of Pericapsular Nerve Group (PENG) Block for Patients Undergoing Shoulder Surgery
Brief Title: Ultrasound-guided PENG Block for Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBFS
Record Dates: First submitted 2021-09-11; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Pain After Shoulder Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Procedure: Pericapsular nerve group block
- Group B (Active Comparator)
  Interventions: Procedure: Interscalene block

INTERVENTIONS:
Procedure: Pericapsular nerve group block — A new nerve block guided by ultrasound that aims to block articular branches of the shoulder.
  Arms: Group A
Procedure: Interscalene block — A common and rapid-onset nerve block method guided by ultrasound for pain control of patients undergoing shoulder surgery.
  Arms: Group B

SUMMARY:
Significant pain after shoulder surgery induce worse experience and may delay recovery of patients undergoing shoulder surgery. Interscalene brachial plexus block (ISB) is a common and rapid-onset procedure for pain control of patients undergoing shoulder surgery. However, the high incidence of adverse events such as hemidiaphragmatic paresis, horner syndrome after interscalene block threatened patients' safety and raised clinicians' concerns on them. Hence, effective analgesia alternatives to interscalene block with less complications are needed.

Recently, pericapsular Nerve Group (PENG) Block, a new technology is reported for block of articular branches of the shoulder and well pericapsular spread around the glenohumeral joint. In this study, we assume that PENG Block may offer a noinferior analgesia and less incidence of nerve block related adverse events compared with ISB.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* 18 years and older
* Shoulder surgery

Exclusion Criteria:

* Severe pulmonary diseas
* Chronic pain disorders
* Infection of shouler skin
* Pregnant women
* Patients allergy to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores | 3 month
  Pain after the shoulder surgery will be measured using an 11-point numerical rating scale (0 = no pain, 10 = worst pain imaginable).

SECONDARY OUTCOMES:
Adverse events | 3 month

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamak Altinpulluk E, Teles AS, Galluccio F, Simon DG, Olea MS, Salazar C, Fajardo Perez M. Pericapsular nerve group block for postoperative shoulder pain: A cadaveric radiological evaluation. J Clin Anesth. 2020 Dec;67:110058. doi: 10.1016/j.jclinane.2020.110058. Epub 2020 Sep 26. No abstract available. PMID 32987232
- [Background] Yamak Altinpulluk E, Galluccio F, Salazar C, Olea MS, Garcia Simon D, Espinoza K, Teles AS, Gonzalez-Arnay E, Fajardo Perez M. A novel technique to Axillary Circumflex Nerve Block: Fajardo approach. J Clin Anesth. 2020 Sep;64:109826. doi: 10.1016/j.jclinane.2020.109826. Epub 2020 Apr 16. No abstract available. PMID 32305791
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Background] Lee MG, Shin YJ, You HS, Lim CH, Chang YJ, Shin HJ. A Comparison of Anesthetic Quality Between Interscalene Block and Superior Trunk Block for Arthroscopic Shoulder Surgery: A Randomized Controlled Trial. Pain Physician. 2021 May;24(3):235-242. PMID 33988942